CLINICAL TRIAL: NCT00176774
Title: A Pilot Trial of Irinotecan, 5-Fluorouracil, and Leucovorin Combined With the Anti-Angiogenesis Agent Tetrathiomolybdate in Metastatic Colorectal Carcinoma (UMCC 0075)
Brief Title: Irinotecan, 5-Fluorouracil, and Leucovorin in Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Dr. Mark Zalupski, University of Michigan Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 0075
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin; tetrathiomolybdate

INTERVENTIONS:
Drug: Irinotecan — Irinotecan by intravenous infusion (needle in a vein in your arm) over 90 minutes immediately followed by intravenous LV and 5-FU weekly for 4 weeks (days 1, 8, 15 and 22) followed by two weeks of no treatment.
Drug: 5-Fluorouracil — Irinotecan by intravenous infusion (needle in a vein in your arm) over 90 minutes immediately followed by intravenous LV and 5-FU weekly for 4 weeks (days 1, 8, 15 and 22) followed by two weeks of no treatment.
Drug: Leucovorin — Irinotecan by intravenous infusion (needle in a vein in your arm) over 90 minutes immediately followed by intravenous LV and 5-FU weekly for 4 weeks (days 1, 8, 15 and 22) followed by two weeks of no treatment.
Drug: Tetrathiomolybdate — one 40 mg oral (by mouth) dose of TM three times a day with meals and one 60 mg oral dose (without food) at bedtime beginning at bedtime on day 1 of your first 6-week cycle of treatment. The between meal dose must be taken at least one hour before or one hour after a meal.

SUMMARY:
This study will examine an investigational (experimental) agent Tetrathiomolybdate (TM) combined with the chemotherapy drugs Irinotecan, 5-Fluorouracil (5-FU) and Leucovorin (LV). This study will evaluate the safety and tolerability of the combination of these drugs when they are used in the treatment of metastatic colorectal cancer.

This is a pilot clinical trial which will be studying the reactions of the patient's body and tumor to the experimental treatment described above. The purpose of this study is to find out what kind of side effects this experimental treatment causes and see how often these side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven adenocarcinoma primary to the colon or rectum and clinical or pathologic evidence of distant metastasis.
* Patients may have received adjuvant chemotherapy and/or one regimen of chemotherapy for metastatic disease. Patients must not have been previously treated with the combination of irinotecan/5-FU/LV.
* Patients must be past their 18th birthday at the time of enrollment.
* Patients must have a performance status of 0-2 at the time of registration.
* Patients must have a life expectancy of > 3 months.
* If patients have undergone recent surgery, they must have fully recovered from the effects of that surgery prior to enrollment.
* Patients must have a pretreatment leukocyte count > 3,000/l, absolute neutrophil count >1500/l, hemoglobin >8 mg/dl, and platelet count of > 150,000/l within 2 weeks of enrollment.
* Patients must have adequate renal function, as documented by a serum creatinine < 2.0 mg/dl, and have adequate hepatic function, as documented by a serum bilirubin < 1.1 mg/dl within 2 weeks of enrollment.

Exclusion Criteria:

* Patients must not have active infection.
* Patients must have no serious medical or psychiatric illness, other than that treated by this study, which would limit the ability of the patient to receive protocol therapy or give informed consent.
* Patients must not have a history of active malignancy, other than that treated by this study, within the 12 months preceding enrollment.
* Pregnant or lactating women may not participate. Women of reproductive age must undergo a serum pregnancy test within 14 days of enrollment. Men and women of reproductive potential must use an effective contraceptive method during the study.
* There must be no plans for the patient to receive concomitant antineoplastic therapy while on this protocol.

All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-02; Primary Completion 2004-02 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
OBJECTIVES | 12 months
To determine the tolerability and toxicity of tetrathiomolybdate (TM) in combination with irinotecan, 5-fluorouracil (5-FU), and leucovorin (LV) in metastatic colorectal cancer. | 12 months
Toxicity | 12 months

SECONDARY OUTCOMES:
To evaluate the progression free survival in patients with metastatic colorectal cancer when treated with this regimen. | 24 months
To determine the tolerability and toxicity of tetrathiomolybdate (TM) in combination with irinotecan, 5-fluorouracil (5-FU), and leucovorin (LV) in metastatic colorectal cancer. | 12 months
To determine the success rate of TM leading to target levels of copper depletion in patients treated concurrently with chemotherapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States